CLINICAL TRIAL: NCT06773559
Title: Comparison of Posture, Balance, Gait and Plantar Pressure Parameters of Transfemoral Amputees in Different Prosthesis Use Periods
Brief Title: Comparison of Transfemoral Amputees in Different Prosthesis Use Periods
Status: Completed | Type: Observational
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Mustafa Sarı, Research Assistant, Lokman Hekim University
Other Study IDs: 2023187
Record Dates: First submitted 2024-11-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Transfemoral Amputees
MeSH Terms: interventions — Gait

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Transfemoral amputee group using prosthesis for at least 3 years
  Interventions: Diagnostic Test: plantar pressure, gait and static balance analysis; Diagnostic Test: trunk posture analysis
- New transfemoral amputee group using prosthesis between two and six weeks
  Interventions: Diagnostic Test: plantar pressure, gait and static balance analysis; Diagnostic Test: trunk posture analysis
- Healthy adult group
  Interventions: Diagnostic Test: plantar pressure, gait and static balance analysis; Diagnostic Test: trunk posture analysis

INTERVENTIONS:
Diagnostic Test: plantar pressure, gait and static balance analysis — Plantar pressure, gait and static balance analysis performed using Ultium Insole SmartLead insoles.
Diagnostic Test: trunk posture analysis — Trunk posture analysis was performed using Diers Formetric 4D.

SUMMARY:
Nowadays, the use of prostheses is recognised as a critical rehabilitation tool for individuals who have experienced limb loss as a result of amputation in order to improve their quality of life and help them return to their activities of daily living. Prostheses offer the potential to help these individuals regain their mobility as well as optimise their physical function. Especially for unilateral transfemoral amputees, there are a number of physical challenges they face during prosthesis use. These challenges can manifest as posture, balance and weight transfer problems that prosthesis users face in their daily lives. Correcting trunk posture, increasing the ability to maintain static balance and optimising plantar load distribution are critical factors affecting the success of prosthesis use. These challenges faced by unilateral transfemoral amputees during prosthesis use are closely related to post-amputation biomechanical changes. These changes can often lead to problems with balance, gait and functionality during activities of daily living. There is no effective comparative study based on computerised analysis data on posture assessment, static balance and plantar pressure distribution of transfemoral amputees.The aim of this study was to investigate the effects of prosthesis use by comparing posture, balance, gait and plantar pressure parameters of unilateral transfemoral amputees at different prosthesis use periods

ELIGIBILITY:
Inclusion Criteria:

* To be using unilateral hydraulic knee joint and carbon foot prosthesis.
* Being amputee at the transfemoral level
* Being new or using prosthesis for at least 3 years.
* Having undergone amputation due to trauma.
* To have completed prosthetic period rehabilitation.
* To be between the ages of 18-45

Exclusion Criteria:

* Having a wound-ulcer problem
* Having amputation due to diabetes, peripheral arterial disease, tumour or venous insufficiency
* Being diagnosed with any systemic or neurological disease
* Affected perception and cognition
* Body mass index above 30.
* Having lower extremity contracture

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteer transfemoral amputees and healthy adults
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Plantar pressure analysis | Baseline
  It was evaluated using the insoles of the Ultium Insole SmartLead. This system is compatible with the Ultium EMG system and can be used in a portable laboratory environment. It is also capable of providing users with zoned and total normalised load-time curves. In addition, it provides users with data such as 3D pressure animations and pressure centre, enabling a more detailed analysis of load distribution. These features make load distribution analysis for clinical or research purposes more effective and user-friendly. It also provides the possibility to monitor relative load distribution during balancing and bilateral or unilateral exercise applications. Applications of this technology include static and dynamic load imbalance detection, and body sway analysis.
Gait analysis | Baseline
  Duration-distance characteristics of gait were evaluated using Ultium Insole SmartLead insoles. This system is compatible with the Ultium EMG system and can be used in a portable laboratory environment. It enables contact detection and quantitative analysis in walking, running and other dynamic activities. Applications of this technology include gait analysis, and running analysis.

SECONDARY OUTCOMES:
Trunk posture analysis | Baseline
  Evaluated with the DIERS Formetric 4D Analysis System. The system offers the ability to perform fast and radiation-free static and dynamic (functional) optical measurements of the human spine. This system works without contact and can objectively analyse spinal posture, scoliosis and other spinal deformities with various clinical parameters.
Fear of falling | Baseline
  It was assessed with the International Falls Efficacy Scale (FES-I): Fear of falling can reduce a person's quality of life and lead to a range of negative consequences, including psychological distress, increased medication use, activity limitations, decreased physical functioning, increased risk of falls, and the need for institutional care. The FES measures confidence in performing activities of daily living without falling. This scale has an excellent performance in terms of reliability and is correlated with balance and gait measures. It is also known for its ability to predict future falls and decline in functional capacity. The FES-I is a scale used to assess fear of falling and was developed as an international version of the Falls Efficacy Scale. The FES-I is used to assess individuals' fear of falling and their confidence in performing daily activities. The FES-I is frequently used by health professionals to determine fear of falling and to assess the need for intervention.
Body image | Baseline
  It was evaluated with the Amputee Body Image Scale (ABIS). The scale is recognised as an important tool in the process of understanding and improving the body image of amputees. It was developed to assess the body experiences of amputees. The ABIS contains 20 items and measures the perceptions and feelings of the person about his/her body after amputation. During its development, important psychometric properties such as content validity, internal consistency and validity were found acceptable.
Satisfaction level | Baseline
  It was evaluated with the Prosthesis Satisfaction Questionnaire. This questionnaire assesses the satisfaction of amputees with their prostheses. The questionnaire consists of 15 questions, and for each question, the participants tick one of the following options: 3: completely agree, 2: strongly agree, 1: disagree, 0: strongly disagree and receive the appropriate score. The total score ranges from 0 to 45, with higher scores indicating higher levels of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Sogutozu, Turkey (Türkiye)